CLINICAL TRIAL: NCT07269145
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of TQB3122 Capsules in Subjects With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3122-I-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3122 Capsules (Experimental): TQB3122 Capsules: Administer once daily, recommended to be taken orally on an empty stomach in the morning at a fixed time, continuously, with each 28-day period as one treatment cycle.
  Interventions: Drug: TQB3122 Capsules

INTERVENTIONS:
Drug: TQB3122 Capsules — TQB3122 Capsules is a poly(ADP - ribose) polymerase 1 (PARP1) -targeted inhibitor.

SUMMARY:
This is the first-in-human clinical study of TQB3122, aiming to evaluate the safety, tolerability, and pharmacokinetic characteristics of TQB3122 in advanced solid tumors, and to preliminarily explore its efficacy in solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily participates in this study, signs the informed consent form, and has good compliance;
* Gender is not restricted; age (calculated as of the date of signing the informed consent form): 18-75 years old;
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0-1; expected survival period ≥ 3 months;
* Patients with histologically or cytologically confirmed advanced malignant solid tumors, including but not limited to epithelial ovarian cancer, fallopian tube cancer, primary peritoneal cancer, breast cancer, prostate cancer, etc.;
* Advanced solid tumors that have failed standard treatment (disease progression or intolerance) or for which there is no standard treatment plan;
* For Phase Ib (dose expansion stage), except for patients receiving maintenance treatment for ovarian cancer/fallopian tube cancer/primary peritoneal cancer, other patients are required to have target lesions meeting the RECIST 1.1 criteria. For Phase Ia (dose escalation stage), measurable lesions are not required;
* Good function of major organs;
* Women of childbearing age must agree to use effective contraceptive measures during the study and within 6 months after the end of the study; serum or urine pregnancy test must be negative within 7 days before enrollment, and they must be non-lactating subjects; men must agree to use effective contraceptive measures during the study and within 6 months after the end of the study.

Exclusion Criteria:

* History of other malignant tumors within 3 years prior to the first administration of the study drug;
* Failure to recover from toxicity and/or complications of previous interventions to CTCAE ≤ Grade 1;
* Risk of bleeding;
* Arterial thrombotic events occurring within 6 months prior to the first administration;
* Suffering from ≥ Grade 2 myocardial ischemia or myocardial infarction, supraventricular or ventricular arrhythmias, and ≥ Grade 2 congestive heart failure; poorly controlled blood pressure;
* History of psychotropic substance abuse with inability to abstain, or presence of mental disorders; patients with epilepsy requiring treatment; or patients with severe mental or neurological diseases;
* Active or uncontrolled severe infections;
* Active syphilis; HIV infection or other immunodeficiency diseases; active hepatitis B or active hepatitis C;
* Complicated with moderate to severe pulmonary diseases that significantly affect respiratory function;
* Patients with active autoimmune diseases requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants);
* Receipt of systemic treatment with prednisone > 10 mg/day or equivalent drugs, or any other form of immunosuppressive therapy within 2 weeks prior to administration;
* History of organ transplantation (except corneal transplantation), allogeneic or autologous hematopoietic stem cell transplantation;
* Poorly controlled diabetes mellitus;
* Patients with leptomeningeal (including arachnoid and pia mater) metastases;
* Known central nervous system (CNS) involvement;
* Presence of massive serous cavity (pleural, peritoneal, or pericardial) effusions requiring repeated drainage to relieve clinical symptoms, or receipt of therapeutic serous cavity effusion drainage within 2 weeks prior to treatment;
* Current intestinal obstruction;
* Known allergy to the components of the study drug;
* Receipt of anti-tumor treatments such as radiotherapy, chemotherapy, targeted therapy, or immunotherapy within 4 weeks prior to the first administration;
* Receipt of Chinese patent medicines explicitly indicated for anti-tumor use in their drug labels approved by National Medical Products Administration (NMPA) within 2 weeks prior to the first administration;
* According to the investigator's judgment, subjects with concomitant diseases that severely endanger their safety or affect the completion of the study, or those deemed unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (each cycle is 28).
  DLT will be defined as toxicities that meet pre-defined severity criteria(according to the NCI Common Terminology Criteria for Adverse Events(CTCAE) version5.0 toxicity assessment criteria), and assessed as having a suspected relationship to study drug that occurred from the first dose to the end of the first treatment cycle.
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 28).
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Recommended Phase II Dose (RP2D) | Baseline up to 24 months
  DLT describes side effects of a drug or other treatment that are serious enough to evaluate RP2D of TQB3122 capsules in adult patients with Breast cancers.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  Defined as the proportion of subjects with complete response (CR), partial response (PR), or Stable Disease (SD).
Overall Survival (OS) | Baseline up to die, estimated one year
  From randomization to the time of death from any cause.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Meizhou People's Hospital (Meizhou Academy of Medical Sciences), Meizhou, Guangdong
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan